CLINICAL TRIAL: NCT04453813
Title: A Multicenter Randomized Clinical Phase 3 Trial of Toripalimab Plus Concurrent Chemo-radiotherapy vs Concurrent Chemo-radiotherapy Alone for Unresectable Locally Recurrent Nasopharyngeal Carcinoma
Brief Title: Toripalimab Plus Concurrent Chemo-radiotherapy for Unresectable Locally Recurrent Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Yuebei People's Hospital (Other); Wuzhou Red Cross Hospital (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Professor, Chief Doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-MYC-2020-2101
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Nasopharyngeal Carcinoma; Chemotherapy; Radiotherapy; PD-1 Treatment
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toripalimab plus concurrent chemo-radiotherapy arm (Experimental): Concurrent chemo-radiotherapy plus concurrent and adjuvant toripalimab.
  Interventions: Drug: Toripalimab plus concurrent chemo-radiotherapy
- Concurrent chemo-radiotherapy arm (Active Comparator): Concurrent chemo-radiotherapy alone.
  Interventions: Drug: Concurrent chemo-radiotherapy

INTERVENTIONS:
Drug: Toripalimab plus concurrent chemo-radiotherapy — 1. Toripalimab: 240 mg, intravenous injection over 60 minutes (Q3W); 2 cycles of toripalimab are concurrently used during radiotherapy and other 9 cycles of toripalimab are used after the end of radiotherapy. (A total of 11 cycles).
  2. Concurrent cisplatin chemotherapy: cisplatin is given at a dose of 100 mg/m2 via a continuous intravenous infusion during radiotherapy and starts on the 1st day of radiotherapy for 2 cycles. 1 cycles per 3 weeks.
  3. IMRT: PTVnx#60.0Gy/27Fr/2.22Gy; PTVnd# 60-64Gy/27Fr/2.22-2.37Gy; PTV1#54Gy/27Fr/2.00Gy
  Arms: Toripalimab plus concurrent chemo-radiotherapy arm
Drug: Concurrent chemo-radiotherapy — 1. Concurrent cisplatin chemotherapy: cisplatin is given at a dose of 100 mg/m2 via a continuous intravenous infusion during radiotherapy and starts on the 1st day of radiotherapy for 2 cycles. 1 cycles per 3 weeks.
  2. IMRT: PTVnx#60.0Gy/27Fr/2.22Gy; PTVnd# 60-64Gy/27Fr/2.22-2.37Gy; PTV1#54Gy/27Fr/2.00Gy
  Arms: Concurrent chemo-radiotherapy arm

SUMMARY:
Through multicenter, open-label, randomised clinical trials, we intend to demonstrate that concurrent and adjuvant PD-1 treatment added to concurrent chemo-radiotherapy could further decrease the rate of disease progression and improve the survival outcome of patients with unresectable locally recurrent nasopharyngeal carcinoma compared with those treated with concurrent chemo-radiotherapy alone.

DETAILED DESCRIPTION:
Through multicenter, open-label, randomised clinical trials, patients with unresectable locally recurrent nasopharyngeal carcinoma are randomized into concurrent chemo-radiotherapy plus concurrent and adjuvant PD-1 treatment group and concurrent chemo-radiotherapy alone group. The efficacy and safety of patients between these two groups are compared.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed recurrent nasopharyngeal carcinoma.
2. The recurrence time is more than 12 months from the end of the first course of radiotherapy.
3. Tumor staged as rT2-4N0-3M0，rII-IVa (according to the 8th AJCC edition).
4. Subjects must have a measurable disease by CT or MRI per RECIST 1.1 criteria.
5. Karnofsky scale (KPS)≥70.
6. Normal bone marrow function.
7. Normal liver and kidney function:

   1. total bilirubin, AST and ALT levels of no more than 2.5 times the upper normal limit;
   2. creatinine clearance rate of at least 60 mL/min or creatinine of no more than 1.5 times the upper normal limit.
8. Given written informed consent.

Exclusion Criteria:

1. Resectable nasopharyngeal diseases: rT2 (the tumour is confined in the superficial parapharyngeal spacer and is more than 0.5cm from the internal carotid artery) and rT3 (the tumour is confined in the base wall of the sphenoid sinus and is more than 0.5cm from the internal carotid artery and cavernous sinus).
2. The patients are suffering from severe nasopharyngeal necrosis, radiation induced brain injury, and fibrosis of the neck et. al, who are evaluated as unsuitable for secondary radiotherapy by the researchers.
3. Has known allergy to large molecule protein products or any compound of study therapy.
4. Has known subjects with other malignant tumors.
5. Has any active autoimmune disease or history of autoimmune disease.
6. Has a history of psychiatric substance abuse, alcoholism, or drug addiction.
7. The laboratory examination value does not meet the relevant standards within 7 days before enrollment
8. Received a systematic glucocorticoid therapy within 4 weeks of the first dose of study medication.
9. Has a known history of active TB (bacillus tuberculosis) within 1 year; patients with adequately treated active TB with 1 year.
10. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or CTLA-4 agent.
11. Has active autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, and asthma requiring bronchodilator therapy). Patients with skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia) will be allowed to enroll.
12. Has a known history of human immunodeficiency virus (HIV).
13. Has hepatitis B surface antigen (HBsAg) positive with HBV DNA copy number of ≥1000cps/ml or hepatitis C virus (HCV) antibody positive
14. Has received a live vaccine within 4 weeks of planned start of study therapy
15. Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 3 years
  Defined as time from randomization to locoregional or distant metastasis relapse or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  Defined as the time interval from randomization to death due to any cause.
Distant Metastasis-Free Survival (DMFS) | 3 years
  Defined as the time interval from randomisation to the date of first distant metastases.
Locoregional Relapse-Free Survival (LRRFS) | 3 years
  Defined as the time from randomisation to the date of first locoregional relapse.
Incidence of treatment related acute complications | up to 1 years
  The proportion of patients with treatment related acute complications according to NCI-CTC5.0 criteria and RTOG criteria.
Incidence of treatment related late complications | up to 3 years
  The proportion of patients with treatment related late complications according to NCI-CTC5.0 criteria and RTOG criteria.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | up to 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | up to 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi